CLINICAL TRIAL: NCT07311681
Title: Break Down the Moves of Laparoscopic Suturing: Stepwise Training Program
Brief Title: Stepwise Versus Conventional Training in Laparoscopic Suturing
Acronym: stepwisetrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Stepwise vs. Conventional
Record Dates: First submitted 2025-12-08; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Learning Outcomes of Laparoscopic Suturing
Keywords: laparoscopic suturing; laparoscopic training; stepwise training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepwise (Experimental): Participants undergoing stepwise training
  Interventions: Other: stepwise training for laparoscopic suturing
- Conventional (Other): Participants undergoing conventional training
  Interventions: Other: conventional training for laparoscopic suturing

INTERVENTIONS:
Other: stepwise training for laparoscopic suturing — Pick up needle: 10 mins (5 mins for each hand) Control needle angle: 20 mins (10 mins for each participant) Needle drive and pull thread: 20 mins (10 mins for each participant) Make double throws: 20 mins (10 mins for each participant) Knot tying: 20 mins (10 mins for each participant) Free practice: 30 mins (15 mins for each participant)
  Arms: Stepwise
Other: conventional training for laparoscopic suturing — Repeating laparoscopic suturing all over
  Arms: Conventional

SUMMARY:
This study will compare the learning outcomes between the participants undergoing stepwise training and conventional training for laparoscopic suturing.

ELIGIBILITY:
Inclusion Criteria:

* the 5th-years medical students in academic year 2020-2021 and 2022-2023

Exclusion Criteria:

* not consenting the research or not completing the training program or tests

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
suturing time | From the first course to the 2nd post-course test in 2 months
  the time to finish a standardized laparoscopic suturing knot
Laparoscopic suturing competency assessment tool | From the first course to the 2nd post-course test in 2 months
  a validated assessment tool for laparoscopic suturing. The lowest score is 8, which represents the best skill level. The high the score is, the poorer the skill level is.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No